CLINICAL TRIAL: NCT01967355
Title: Prolongation of Pregnancy in Preeclampsia by Therapeutic Lipid Apheresis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karl Winkler (Other)
Responsible Party: Sponsor-Investigator, Karl Winkler, Professor Dr. med., University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-15
Record Dates: First submitted 2013-07-26; First posted 2013-10-22 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Preeclampsia; Dyslipidemia; Proteinuria; Hypertension
Keywords: preeclampsia; lipid apheresis; apheresis
MeSH Terms: conditions — Pre-Eclampsia; Dyslipidemias; Proteinuria; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lipid apheresis (Experimental): Lipid apheresis: lipid removing therapy,frequency and duration depending on the symptoms of mother and fetus.
  Interventions: Other: lipid apheresis

INTERVENTIONS:
Other: lipid apheresis
  Other Names: H.E.L.P.-Apheresis

SUMMARY:
Preeclampsia is a disease which occurs in about 6-8% of all pregnancies and is the main cause of maternal and fetal morbidity and mortality. The cause of preeclampsia is still not clear and the only therapy is preterm caesarean section. In severe preeclampsia an accumulation of triglyceride-rich lipoproteins occurs. Therefore, lipid apheresis is performed as lipid-removing therapy for treatment of preeclampsia in order to prolong pregnancy and provide the fetus more time for maturation. In this individual treatment patients with early preeclampsia (<= 32 weeks of gestation) will be offered a H.E.L.P.-apheresis to postpone caesarean section and therefore prolong pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* early preeclampsia (< 32 week of pregnancy)
* arterial hypertension during pregnancy
* proteinuria (=> 1 + dipstick or 0> 300 mg/24h)
* and/or intrauterine growth retardation (IUGR)
* informed consent

Exclusion Criteria:

* every acute indication for immediate delivery
* no informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-04; Primary Completion 2014-05-08 (Actual); Study Completion 2014-05-08 (Actual)

PRIMARY OUTCOMES:
Prolongation of pregnancy | Mother will be followed up for the duration of hospital stay, that is from first lipid apheresis until the discharge of the mother in the days following birth (an expected average of 3-4 weeks).
  A deteriorating clinical condition of the mother and the fetus necessitates a caesarean section (c.s.). However, if c.s. takes place too early lung maturation of the fetus may not be completed. Apheresis is initiated and will be continued until lung maturity is achieved and the clinical condition of the mother and the fetus improves.

SECONDARY OUTCOMES:
Reduction of lipoprotein levels | Mother will be followed up for the duration of hospital stay, that is from first lipid apheresis until the discharge of the mother in the days following birth (an expected average of 3-4 weeks).

OTHER OUTCOMES:
Normalization of blood pressure measured in mmHg. | Mother will be followed up for the duration of hospital stay, that is from first lipid apheresis until the discharge of the mother in the days following birth (an expected average of 3-4 weeks).
Normalization of proteinuria measured in 24-h urine collection in mg/dl | Mother will be followed up for the duration of hospital stay, that is from first lipid apheresis until the discharge of the mother in the days following birth (an expected average of 3-4 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Karl Winkler, Prof.Dr.med., Principal Investigator — Institute of Clinical Chemestry and Laboratory Medicine, University Hospital Freiburg
Locations (1):
- Institute of Clinical Chemistry and Laboratory Medicine, University Hospital Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Winkler K, Lorey C, Contini C, Augustinski V, Putz G, Rothele E, Benner A, Fuchs H, Pecks U, Markfeld-Erol F, Kunze M. Comparison of double-filtration plasmapheresis (DFPP) versus heparin-mediated extracorporeal LDL-precipitation (HELP)-apheresis in early-onset preeclampsia. Pregnancy Hypertens. 2024 Jun;36:101128. doi: 10.1016/j.preghy.2024.101128. Epub 2024 May 9. PMID 38728925
- [Derived] Contini C, Jansen M, Konig B, Markfeld-Erol F, Kunze M, Zschiedrich S, Massing U, Merfort I, Prompeler H, Pecks U, Winkler K, Putz G. Lipoprotein turnover and possible remnant accumulation in preeclampsia: insights from the Freiburg Preeclampsia H.E.L.P.-apheresis study. Lipids Health Dis. 2018 Mar 14;17(1):49. doi: 10.1186/s12944-018-0698-4. PMID 29540222